CLINICAL TRIAL: NCT00192595
Title: Virological and Clinical Anti-HBV Efficacy of Tenofovir in Antiretroviral naïve Patients With HIV/HBV Co-infection
Brief Title: Tenofovir in HIV/HBV Coinfection
Acronym: TICO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); Gilead Sciences (Industry)
Responsible Party: A/Prof Gregory J Dore, National Centre in HIV Epidemiology and Clinical Research, Univeristy of New South Wales
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHWG001; TICO
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection; Hepatitis B Coinfection
Keywords: Hepatitis B; HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Tenofovir; Zidovudine; Lamivudine; lipoarabinomannan; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: (Active Comparator): Zidovudine (AZT), lamivudine (LAM), efavirenz (EFV)
  Interventions: Drug: Zidovudine (AZT), lamivudine (LAM), efavirenz (EFV)
- Arm 2 (Experimental): Zidovudine (AZT), tenofovir (TDF), efavirenz (EFV)
  Interventions: Drug: Tenofovir
- Amr 3 (Experimental): Lamivudine (LAM), tenofovir (TDF), efavirenz (EFV)
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir
  Arms: Amr 3; Arm 2
Drug: Zidovudine (AZT), lamivudine (LAM), efavirenz (EFV)
  Arms: Arm 1:

SUMMARY:
The purpose of the study is to compare the effectiveness of 3 different treatment regimens in reducing or clearing the Hepatitis B Virus in patients infected with HIV and Hepatitis B (co-infection)

DETAILED DESCRIPTION:
A randomised multi-centre trial of tenofovir vs lamivudine vs tenofovir/lamivudine in antiretroviral naïve subjects with HIV/HBV co-infection over 48 weeks (Clinical Trial A). Plus, a 12 week viral kinetic sub-study comparing a sub-group of the patients on Clinical Trial A with a group of therapy naïve HBV mono-infected subjects (Substudy A1)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Documented HIV infection (positive serology for HIV-1 and detectable HIV-1 RNA)
* Age 18 - 70 years
* HBV DNA > 105 copies/ml
* HBsAg positive >6 months or HBsAg positive and anti HB core IgM negative
* Creatinine <= 2.0mg/dl (<= 0.2 mmol/L)
* Platelet count >= 50,000/mm
* HIV-1 antiretroviral therapy naïve
* No prior exposure to anti-HBV agents (LAM, adefovir, TDF) although prior IFN treatment allowed

Exclusion Criteria:

* HCV-RNA positive or Anti-HAV IgM positive
* Acute hepatitis (serum ALT > 1000 U/L)
* Active opportunistic infection
* Other causes of chronic liver disease identified (autoimmune hepatitis, hemochromatosis, Wilsons disease, alfa-1-antitrypsin deficiency)
* Concurrent malignancy requiring cytotoxic chemotherapy
* Decompensated or Child's C cirrhosis
* Alfa-fetoprotein (AFP) > 3X ULN (unless negative CT scan or MRI within 3 months of entry date)
* Pregnancy or lactation
* Any other condition which in the opinion of the investigator might interfere with compliance or outcome of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To compare HBV DNA suppression to levels below the limit of detection (<400 copies/ml) by week 48 in each group

SECONDARY OUTCOMES:
-HBV resistance at 48 weeks; -undetectable HBV DNA at weeks 12 & 24; -HBeAg and HBsAg seroconversion at weeks 24 & 48; -ALT chnages and rate of hepatic cytolysis; -HIV-1 RNA supression and CD4/CD8 changes over 48 weeks;

CONTACTS AND LOCATIONS:
Overall Officials: Greg Dore, MBBS, FRACP, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.
Locations (3):
- Australia (2):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand

REFERENCES:
- [Derived] Avihingsanon A, Matthews GV, Lewin SR, Marks P, Sasadeusz J, Cooper DA, Bowden S, Locarnini S, Dore GJ, Ruxrungtham K. Assessment of HBV flare in a randomized clinical trial in HIV/HBV coinfected subjects initiating HBV-active antiretroviral therapy in Thailand. AIDS Res Ther. 2012 Mar 9;9(1):6. doi: 10.1186/1742-6405-9-6. PMID 22405335
- [Derived] Matthews GV, Avihingsanon A, Lewin SR, Amin J, Rerknimitr R, Petcharapirat P, Marks P, Sasadeusz J, Cooper DA, Bowden S, Locarnini S, Ruxrungtham K, Dore GJ. A randomized trial of combination hepatitis B therapy in HIV/HBV coinfected antiretroviral naive individuals in Thailand. Hepatology. 2008 Oct;48(4):1062-9. doi: 10.1002/hep.22462. PMID 18697216
- See also: National Centre in HIV Epidemiology and Clinical Research — http://www.med.unsw.edu.au/nchecr